CLINICAL TRIAL: NCT04016311
Title: A Brief Mindful Drinking/Eating Intervention for Hemodialysis Patients With Fluid Restrictions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Gayle Timmerman,, Associate Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-01-0074
Record Dates: First submitted 2019-07-08; First posted 2019-07-11 (Actual); Results first posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Kidney Failure; Quality of Life; Fluid Restriction; Interdialytic Weight Gain; Hemodialysis; Mindfulness
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Intervention and wait list control groups with rolling admission.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Drinking/Eating Group (Experimental): Behavioral: Mindful Drinking/Eating Intervention Participants will be individually guided during their dialysis session through: 1) a mindful drinking exercise, a meditation focused on the sensory experience of 3 sips of fluid, along with a discussion of the experience; and 2) a mindful eating exercise with select foods that are recommended for controlling thirst (i.e., hard candy, frozen fruits). Participants will be given directions for mindful drinking/eating and asked to practice mindful drinking/eating as often as possible but least once each day.
  Interventions: Behavioral: Mindful Drinking/Eating Intervention
- Wait list control (No Intervention): Usual care. Offered intervention after post-test data collected.

INTERVENTIONS:
Behavioral: Mindful Drinking/Eating Intervention — Participants will be individually guided during their dialysis session through: 1) a mindful drinking exercise, a meditation focused on the sensory experience of 3 sips of fluid, along with a discussion of the experience; and 2) a mindful eating exercise with select foods that are recommended for controlling thirst (i.e., hard candy, frozen fruits). Participants will be given directions for mindful drinking/eating and asked to practice mindful drinking/eating as often as possible but least once each day.
  Arms: Mindful Drinking/Eating Group

SUMMARY:
The purpose of this pilot study is to find out whether mindful drinking/eating activities can improve quality of life and help make it easier for people on dialysis to follow their fluid restrictions. The pilot study is a randomized controlled trial with an intervention group and a wait list control group, randomized by cohort days. The intervention occurs during dialysis sessions once a week for 4 weeks. During each intervention session, participants are guided through a mindful eating exercise focused on foods recommended for controlling thirst (e.g., hard candy, frozen grapes) and a mindful drinking exercise. Participants are asked to practice mindful drinking/eating at least once daily at home.

ELIGIBILITY:
Inclusion Criteria:

* Receiving hemodialysis
* Able to speak English

Exclusion Criteria:

* Missed more than one dialysis treatment in the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from 2 dialysis centers. Assigned randomly by cohort (Tues/Thurs/Sat dialysis patients vs Monday/Wed/Friday) to prevent contamination.
Groups:
- Wait List Control: Usual treatment - offered intervention after completion of post-test data collection.
Period: Overall Study
Arm/Group | Mindful Drinking/Eating Group | Wait List Control
Started | 18 | 20
Completed | 17 | 20
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindful Drinking/Eating Group | Wait List Control | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 9 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.56 (13.85) | 61.50 (15.44) | 61.53 (14.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 18
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 7 | 6 | 13
  White | 9 | 12 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 18 | 20 | 38
Total score Kidney Disease Quality of Life -36 SF [Mean (Standard Deviation); unit: units on a scale] — Population: Baseline for study measures does not include the participant that withdrew
  units on a scale
    number analyzed (Participants) | 17 | 20 | 37
    (all) | 68.64 (15.12) | 63.92 (14.91) | 66.09 (14.99)
Interdialytic Weight Gain [Mean (Standard Deviation); unit: kilograms] — Population: Baseline data was analyzed without the data from the participant that withdrew.
  kilograms
    number analyzed (Participants) | 17 | 20 | 37
    (all) | 2.46 (1.10) | 2.52 (1.10) | 2.49 (1.07)
Mindful Eating Questionnaire [Mean (Standard Deviation); unit: units on a scale] — Population: Baseline measure was analyzed without data from the subject that withdrew.
  units on a scale
    number analyzed (Participants) | 17 | 20 | 37
    (all) | 3.08 (0.32) | 2.94 (0.23) | 3.00 (0.28)

OUTCOME MEASURES:

1. Primary Outcome: Total Score for Kidney-Disease Quality of Life Short Form v1.3
Description: Total Score for Kidney-Disease Quality of Life Short Form v1.3 Higher scores indicate greater quality of life. Score range from 0 to 100
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindful Drinking/Eating Group | Wait List Control
Number analyzed (Participants) | 18 | 20
score on a scale | 69.66 (15.79) | 66.12 (13.24)

2. Primary Outcome: Interdialytic Weight Gain (IWG)
Description: Average of 3 Interdialytic Weight gain measures taken the week after last intervention section (4 week time frame). Interdialytic weight gain is calculated as the patients' weight at the beginning of each hemodialysis session (pre-weight) minus the weight after the previous hemodialysis session (post-weight).
  Measured in kilograms. Lower numbers are better. Proxy measure for adhering to fluid restriction.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Mindful Drinking/Eating Group | Wait List Control
Number analyzed (Participants) | 17 | 20
kilograms | 2.86 (1.51) | 2.46 (0.97)

3. Secondary Outcome: Mindful Eating
Description: Total score on Mindful Eating Questionnaire Total Scores range from 1 to 4. Higher scores indicate more mindful eating.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindful Drinking/Eating Group | Wait List Control
Number analyzed (Participants) | 17 | 20
score on a scale | 3.12 (0.26) | 3.03 (0.30)

ADVERSE EVENTS:
Time Frame: Adverse events were tracked from pre-test to post-test per participant over the 4 weeks that they were enrolled in study.
Groups:
- Wait List Control: Usual care. Intervention offered after post-test data collected.
Arm/Group | Mindful Drinking/Eating Group | Wait List Control
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/18 | 2/20
Other Adverse Events (participants affected / at risk) | 0/18 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindful Drinking/Eating Group (N=18) | Wait List Control (N=20)
Hospitalized for fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hospitalized for surgery (Surgical and medical procedures) | 0 (0) | 1 (1) — Pacemaker and Heart valve replacement surgery
Blood clot (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT04016311/Prot_SAP_000.pdf